CLINICAL TRIAL: NCT03090100
Title: A Phase 3, Multicenter, Randomized, Double-blind Study Evaluating the Comparative Efficacy of CNTO 1959 (Guselkumab) and Secukinumab for the Treatment of Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study to Evaluate the Comparative Efficacy of CNTO 1959 (Guselkumab) and Secukinumab for the Treatment of Moderate to Severe Plaque-type Psoriasis
Acronym: ECLIPSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108278; 2016-002995-29 (EudraCT Number); CNTO1959PSO3009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-03-22; First posted 2017-03-24 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I: Guselkumab Plus Placebo (Experimental): Participants will receive 1 injection of active guselkumab and 1 injection of placebo when guselkumab is scheduled to be administered (Weeks 0, 4, 12, 20, 28, 36, and 44) or 2 injections of placebo when no guselkumab is scheduled to be administered (Weeks 1, 2, 3, 8, 16, 24, 32, and 40). Placebo injections will be administered to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group II: Secukinumab (Active Comparator): Participants will receive 2 injections of active secukinumab subcutaneously (SC) at Weeks 0, 1, 2, 3, 4 and every 4 weeks (q4w) thereafter through Week 44.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 1 injection of active guselkumab at Weeks 0, 4, 12, 20, 28, 36, and 44.
  Arms: Group I: Guselkumab Plus Placebo
Drug: Placebo — Participants will receive 1 injection of placebo at Weeks 0, 4, 12, 20, 28, 36, and 44 and 2 injections of placebo at Weeks 1, 2, 3, 8, 16, 24, 32, and 40.
  Arms: Group I: Guselkumab Plus Placebo
Drug: Secukinumab — Participants will receive 2 injections of active secukinumab at Weeks 0, 1, 2, 3, 4 and every 4 weeks (q4w) thereafter through Week 44.
  Other Names: Cosentyx
  Arms: Group II: Secukinumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab compared with secukinumab for the treatment of participants with moderate to severe plaque-type psoriasis.

DETAILED DESCRIPTION:
The study consists of Screening Phase(4 weeks before administration of study drug),Active Treatment Phase(Week 0-Week 44),Follow Up Phase(Week 44-Week 56).During various study periods,safety assessments(example[e.g] recording of adverse events,Vital signs,Tuberculosis evaluation,Chest radiograph,Urine pregnancy Test);Efficacy assessments(e.g IGA,PASI);Clinical Laboratory Assessments(e.g haematology,chemistry);Biomarkers/Genetic evaluations,will be performed per the study procedures.The primary hypotheses are that guselkumab treatment is non-inferior to secukinumab as assessed by proportion of participants achieving PASI 90 response at Week 48 with noninferiority margin of 10% and,once non-inferiority is established,that guselkumab is superior to secukinumab as assessed by proportion of participants achieving PASI 90 response at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis (with or without [Psoriatic Arthritis]PsA) for at least 6 months before the first administration of study drug
* A woman of childbearing potential must have a negative urine pregnancy test at screening and at Week 0 and agree to urine pregnancy testing before receiving injections
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 3 months after the last administration of study drug
* Agree not to receive a Bacille Calmette-Guérin (BCG) vaccination during the study, or within 12 months after the last administration of study drug
* Agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during study

Exclusion Criteria:

* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has previously received guselkumab or secukinumab
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (example bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), fungal infection (mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers
* Has a history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance; or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly
* Is unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (142):
- United States (44):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Southern California Permanente Medical Group, Los Angeles, California
  - Dermatology Specialists, Oceanside, California
  - MedDerm Associates, San Diego, California
  - San Luis Dermatology & Laser Clinic, Inc, San Luis Obispo, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Olympian Clinical Research, Clearwater, Florida
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Renstar Medical Research, Ocala, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia
  - Advanced Medical Research, Atlanta, Georgia
  - Marietta Dermatology Clinical Research, Marietta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Northshore Universite Healthsystem, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - DermAssociates, PC, Rockville, Maryland
  - Great Lakes Research Group, Bay City, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology, St Louis, Missouri
  - Windsor Dermatology, East Windsor, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Dermatologists of Greater Columbus, Bexley, Ohio
  - The Ohio State University, Gahanna, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Austin Dermatology Associates, Austin, Texas
  - Modern Research Associates, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Suzanne Bruce and Associates - The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
- Australia (11):
  - The Skin Centre, Benowa
  - Sinclair Dermatology, East Melbourne
  - Fremantle Dermatology, Fremantle
  - Clinical Trials SA Pty Ltd, Hectorville
  - Premier Specialists, Kogarah
  - St George Dermatology & Skin Cancer Centre, Kogarah
  - Skin&Cancer Foundation Inc, Melbourne
  - Royal Melbourne Hospital, Parkville
  - Westmead Hospital, Westmead
  - Woden Dermatology, Woden
  - Veracity Clinical Research, Woolloongabba
- Canada (14):
  - Dermatrials Research, Hamilton, Ontario
  - Guenther Dermatology Research Centre, London, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - CCA Medical Research Corporation, Ajax
  - Stratica Medical, Edmonton
  - Eastern Canada Research Associates, Halifax
  - DermEdge Research, Mississauga
  - Innovaderm Research, Montreal
  - Centre Dermatologique, Québec
  - Dr. Chih-ho Hong Medical, Surrey
  - K. Papp Clinical Research, Waterloo
  - XLR8 Medical Research, Windsor
- Czechia (8):
  - Nemocnice Jihlava, Jihlava
  - Kozni ambulance Kutna Hora, s.r.o., Kutná Hora
  - DERMAMEDICA s.r.o., Náchod
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - Fakultni nemocnice Ostrava, Ostrava- Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Dermatologicka ambulance, Svitavy
  - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- France (8):
  - CHU Bordeaux - Hopital St Andre, Bordeaux
  - ICH Hopital A. Morvan, Brest
  - Groupe Hospitalier La Rochelle - Re - Aunis, La Rochelle
  - Le Bateau Blanc, Martigues
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Charles Nicolle, Rouen
  - Hopital Larrey CHU de Toulouse, Toulouse
- Germany (17):
  - Charite Universitatsmedizin Berlin, Campus Mitte (CCM) Allergie Center, Berlin
  - ISA GmbH, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Klinische Forschung Dresden GmbH, Dresden
  - University Hospital Dresden, Dresden
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg
  - SCIderm GmbH, Hamburg
  - MensingDerma research GmbH, Hamburg
  - Universitatsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsklinik Luebeck, Lübeck
  - Hautarztpraxis, Mahlow
  - Technische Universitaet Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinik Tuebingen, Tübingen
  - Centrovital, Witten
- Hungary (9):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mor Oktatokorhaz, Kaposvár
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Medmare Egeszsegugyi Es Szolgaltato Bt., Veszprém
- Poland (16):
  - NZOZ Osteo-Medic S.C. Artur Racewicz i Jerzy Supronik, Bialystok
  - Specderm Poznańska sp. j., Bialystok
  - Szpital Uniwersytecki nr 1 im. Dr A. Jurasza, Bydgoszcz
  - Centrum Kliniczno Badawcze, Elblag
  - Copernicus Podmiot Leczniczy Sp. z o.o, Gdansk
  - Malopolskie Centrum Medyczne, Krakow
  - Centrum Badawcze Wspolczesnej Terapii, Lodz
  - Dermed Centrum Medyczne Sp. z o.o, Lodz
  - Solumed S.C., Poznan
  - CRC Sp. z o.o., Poznan
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - NZOZ Poradnia Dermatologiczno-Wenerologiczna Mediderm, Torun
  - Przychodnia Specjalistyczna High-Med, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - DermMedica Sp. z o.o., Wroclaw
  - Centrum Medyczne WroMedica, Wroclaw
- Spain (15):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. de Basurto, Bilbao Vizcaya
  - Hosp. Reina Sofia, Córdoba
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. de Torrejon, Madrid
  - Hosp. de Manises, Manises
  - Hosp. Provincial de Pontevedra, Pontevedra
  - Hosp. Univ. I Politecni La Fe, Valencia

REFERENCES:
- [Derived] Blauvelt A, Chen Y, Branigan PJ, Liu X, DePrimo S, Keyes BE, Leung M, Fakharzadeh S, Yang YW, Munoz-Elias EJ, Krueger JG, Langley RG. Differential Pharmacodynamic Effects on Psoriatic Biomarkers by Guselkumab Versus Secukinumab Correlate with Long-Term Efficacy: An ECLIPSE Substudy. JID Innov. 2024 Jun 26;4(5):100297. doi: 10.1016/j.xjidi.2024.100297. eCollection 2024 Sep. PMID 39224116
- [Derived] Egeberg A, Conrad C, Gorecki P, Wegner S, Buyze J, Acciarri L, Thaci D. Response Types and Factors Associated with Response Types to Biologic Therapies in Patients with Moderate-to-Severe Plaque Psoriasis from Two Randomized Clinical Trials. Dermatol Ther (Heidelb). 2024 Mar;14(3):745-758. doi: 10.1007/s13555-024-01123-1. Epub 2024 Mar 15. PMID 38485863
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Reich K, Armstrong AW, Langley RG, Flavin S, Randazzo B, Li S, Hsu MC, Branigan P, Blauvelt A. Guselkumab versus secukinumab for the treatment of moderate-to-severe psoriasis (ECLIPSE): results from a phase 3, randomised controlled trial. Lancet. 2019 Sep 7;394(10201):831-839. doi: 10.1016/S0140-6736(19)31773-8. Epub 2019 Aug 8. PMID 31402114

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of total 1,048 randomized participants, 534 were assigned to receive Guselkumab + Placebo and 514 subjects were assigned to receive Secukinumab.
Groups:
- Guselkumab 100 mg + Placebo: Participants received 1 injection of active guselkumab and 1 injection of placebo when guselkumab is scheduled to be administered (Weeks 0, 4, 12, 20, 28, 36, and 44) or 2 injections of placebo when no guselkumab is scheduled to be administered (Weeks 1, 2, 3, 8, 16, 24, 32, and 40). Placebo injections were administered to maintain the blind. Participants were continued to follow-up period from Week 44 through Week 56.
- Secukinumab 300 mg: Participants received 2 injections of active secukinumab subcutaneously (SC) at Weeks 0, 1, 2, 3, 4 and every 4 weeks (q4w) thereafter through Week 44. Participants were continued to follow-up period from Week 44 through Week 56.
Period: Overall Study
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Started | 534 | 514
Treated | 534 | 511
Completed | 507 | 466
Not Completed | 27 | 48
Not completed — Adverse Event | 9 | 11
Not completed — Pregnancy | 1 | 1
Not completed — Lack of Efficacy | 2 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 7 | 19
Not completed — Protocol Violation | 2 | 6
Not completed — Non-compliance | 2 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants randomized at Week 0.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg | Total
Number analyzed (Participants) | 534 | 514 | 1048
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 2 | 8
  Between 18 and 65 years | 474 | 467 | 941
  >=65 years | 54 | 45 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.67) | 45.3 (13.57) | 45.8 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 172 | 341
  Male | 365 | 342 | 707
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 36 | 63
  Not Hispanic or Latino | 502 | 472 | 974
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 18 | 12 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 5 | 11 | 16
  White | 499 | 480 | 979
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 35 | 36 | 71
  CANADA | 81 | 77 | 158
  CZECH REPUBLIC | 27 | 28 | 55
  FRANCE | 28 | 30 | 58
  GERMANY | 66 | 56 | 122
  HUNGARY | 25 | 20 | 45
  POLAND | 119 | 119 | 238
  SPAIN | 35 | 33 | 68
  UNITED STATES | 118 | 115 | 233

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI)-90 Response at Week 48
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 48
Population: FAS population included. Participants who met treatment failure criteria (who discontinued study agent due to lack of efficacy or adverse event of psoriasis and/or who initiated protocol-prohibited psoriasis medications/therapies) prior to Week 48 or who had a missing PASI score at Week 48 were considered PASI 90 non-responders at Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 84.5 | 70.0
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Non-Inferiority — Non-inferiority margin of 10%; p < 0.001, z-test; Difference in percentage = 14.2, 95% CI 2-sided [9.2 to 19.2]
Statistical Analysis 2: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants Who Achieved a PASI-75 Response at Both Week 12 and 48
Description: Percentage of participants who achieved PASI-75 response at both Week 12 and 48 was reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 75 response was defined as at least a 75% reduction in PASI relative to baseline.
Time Frame: Week 12 and 48
Population: FAS population included. Participants who met treatment failure criteria (who discontinued study agent due to lack of efficacy or adverse event of psoriasis and/or who initiated protocol-prohibited psoriasis medications/therapies) prior to Week 48 or who had a missing PASI score at Week 12 or 48 were considered as non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 84.6 | 80.2
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Non-Inferiority — Non-inferiority margin of 10%; p < 0.001, z-test; Difference in percentage = 4.3, 95% CI 2-sided [-0.2 to 8.9]
Statistical Analysis 2: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Superiority; p = 0.062, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants Who Achieved a PASI-90 Response at Week 12
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 90 response was defined as at least a 90% reduction in PASI relative to baseline. Due to failing to achieve superiority of prior secondary endpoint, no formal statistical testing was performed for endpoints from this point onwards.
Time Frame: Week 12
Population: FAS population included. Participants who met treatment failure criteria prior to Week 12, who had a missing PASI score at Week 12 were considered PASI 90 non-responders at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 69.1 | 76.1
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -7.0, 95% CI 2-sided [-12.2 to -1.7]

4. Secondary Outcome: Percentage of Participants Who Achieved a PASI-75 Response at Week 12
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 75 response was defined as at least a 75% reduction in PASI relative to baseline.
Time Frame: Week 12
Population: FAS population included. Participants who met treatment failure criteria prior to Week 12 or who had a missing PASI score at Week 12 were considered PASI 75 non-responders at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 89.3 | 91.6
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -2.3, 95% CI 2-sided [-6.0 to 1.2]

5. Secondary Outcome: Percentage of Participants Who Achieved a PASI-100 Response at Week 48
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 100 response was defined as 100% reduction in PASI relative to baseline.
Time Frame: Week 48
Population: FAS population included. Participants who met treatment failure criteria prior to Week 48 or who had a missing PASI score at Week 48 were considered PASI 100 non-responders at Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 58.2 | 48.4
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = 9.7, 95% CI 2-sided [3.8 to 15.5]

6. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score Cleared (0) at Week 48
Description: The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 48
Population: FAS population included. Participants who met treatment failure criteria prior to Week 48 or who had a missing IGA score at Week 48 were considered IGA cleared (0) non-responders at Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 62.2 | 50.4
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = 11.6, 95% CI 2-sided [5.8 to 17.4]

7. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score Cleared (0) or Minimal (1) at Week 48
Description: as for outcome 6
Time Frame: Week 48
Population: FAS population included. Participants who met treatment failure criteria prior to Week 48 or who had a missing IGA score at Week 48 were considered IGA cleared (0) or minimal (1) non-responders at Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 85.0 | 74.9
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = 9.7, 95% CI 2-sided [4.9 to 14.5]

8. Secondary Outcome: Percentage of Participants Who Achieved a PASI-90 Response at Both Week 16 and 48
Description: Percentage of participants who achieved PASI-90 response at both Week 16 and 48 was reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 90 response was defined as at least a 90% reduction in PASI relative to baseline.
Time Frame: Week 16 and 48
Population: FAS population included. Participants who met treatment failure criteria prior to Week 48 or who had a missing PASI score at Week 16 or 48 were considered as non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 72.3 | 64.4
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = 7.8, 95% CI 2-sided [2.3 to 13.2]

9. Secondary Outcome: Percentage of Participants Who Achieved a PASI-75 Response at Week 16
Description: as for outcome 4
Time Frame: Week 16
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria prior to Week 16 or who had a missing PASI score at Week 16 were considered PASI 75 non-responders at Week 16.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 92.7 | 92.8
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -0.3, 95% CI 2-sided [-3.5 to 3.1]

10. Secondary Outcome: Percentage of Participants Who Achieved a PASI-90 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 90 response was defined as at least a 90% reduction in PASI relative to baseline.
Time Frame: Week 16
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria prior to Week 16 or who had a missing PASI score at Week 16 were considered PASI 90 non-responders at Week 16.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 78.5 | 79.6
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -1.4, 95% CI 2-sided [-6.2 to 3.4]

11. Secondary Outcome: Percentage of Participants Who Achieved a PASI-90 Response at All 7 Visits From Week 24 Through Week 48
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 90 response was defined as at least a 90% reduction in PASI relative to baseline. Percentage of participants who achieved a PASI-90 response at all 7 visits from Week 24 to 48 (Week 24, 28, 32, 36, 40, 44 and 48) was reported.
Time Frame: Week 24 up to Week 48
Population: FAS population included. Participants who met treatment failure criteria prior to Week 48 or who had missing PASI score at any visit from Week 24 through 48 were considered as non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 71.0 | 61.5
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = 9.8, 95% CI 2-sided [4.2 to 15.3]

12. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score Cleared (0) or Minimal (1) at Week 16
Description: as for outcome 6
Time Frame: Week 16
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria prior to Week 16 or who had a missing IGA score at Week 16 were considered non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 86.7 | 86.6
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -0.1, 95% CI 2-sided [-4.2 to 3.9]

13. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score Cleared (0) or Minimal (1) at Week 12
Description: as for outcome 6
Time Frame: Week 12
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria prior to Week 12 or who had a missing IGA score at Week 12 were considered non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants | 85.6 | 86.4
Statistical Analysis 1: Comparison: Guselkumab 100 mg + Placebo vs Secukinumab 300 mg; Test type: Other; Difference in percentage = -0.9, 95% CI 2-sided [-5.0 to 3.3]

14. Secondary Outcome: Percentage of Participants Who Achieved PASI-75 Response at Week 48 Among PASI-75 Responders at Week 12
Description: as for outcome 4
Time Frame: Week 48
Population: Full analysis set included all the participants randomized at Week 0 and who achieved PASI 75 response at Week 12. Participants who met treatment failure criteria prior to Week 48 or who had missing PASI score at Week 48 were considered as non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 477 | 471
Percentage of participants | 94.8 | 87.5

15. Secondary Outcome: Percentage of Participants Who Achieved PASI-90 Response at Week 48 Among PASI-90 Responders at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. PASI 90 response was defined as at least a 90 percent (%) reduction in PASI relative to baseline.
Time Frame: Week 48
Population: Full analysis set included all the participants randomized at Week 0 and who achieved PASI-90 response at Week 16. Participants who met treatment failure criteria prior to Week 48 or who had missing PASI score at Week 48 were considered as non-responders for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 419 | 409
Percentage of participants | 92.1 | 80.9

16. Secondary Outcome: Percentage of Participants Who Achieved PASI Response (PASI 100, PASI-90, PASI-75 and PASI-50) Over Time From Week 1 to Week 56
Description: PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body is divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. PASI produces a numeric score that can range from 0 (no psoriasis) to 72.Participants with >=50%, >= 75%, >=90% and 100% improvement in PASI from baseline were considered PASI 50, 75, 90 and PASI 100 responders, respectively.
Time Frame: Week 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 56
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria or who had missing PASI score were considered as non-responders for the specific visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants
  Week 1: 100% improvement | 0 | 0
  Week 1: >=90% improvement | 0 | 0
  Week 1: >=75% improvement | 2.1 | 1.8
  Week 1: >=50% improvement | 10.7 | 12.8
  Week 2: 100% improvement | 0.2 | 0.6
  Week 2: >=90% improvement | 1.1 | 2.7
  Week 2: >=75% improvement | 6.4 | 11.5
  Week 2: >=50% improvement | 30.9 | 42.0
  Week 3: 100% improvement | 1.7 | 1.6
  Week 3: >=90% improvement | 5.6 | 8.6
  Week 3: >=75% improvement | 19.5 | 28.4
  Week 3: >=50% improvement | 56.4 | 66.9
  Week 4: 100% improvement | 4.1 | 5.1
  Week 4: >=90% improvement | 13.1 | 21.8
  Week 4: >=75% improvement | 39.3 | 50.2
  Week 4: >=50% improvement | 73.4 | 85.4
  Week 8: 100% improvement | 20.0 | 27.2
  Week 8: >=90% improvement | 48.7 | 62.1
  Week 8: >=75% improvement | 76.4 | 86.2
  Week 8: >=50% improvement | 95.3 | 96.9
  Week 12: 100% improvement | 37.8 | 42.0
  Week 12: >=90% improvement | 69.1 | 76.1
  Week 12: >=75% improvement | 89.3 | 91.6
  Week 12: >=50% improvement | 96.8 | 96.1
  Week 16: 100% improvement | 47.8 | 46.1
  Week 16: >=90% improvement | 78.5 | 79.6
  Week 16: >=75% improvement | 92.7 | 92.8
  Week 16: >=50% improvement | 97.6 | 96.3
  Week 20: 100% improvement | 51.3 | 48.6
  Week 20: >=90% improvement | 80.1 | 81.1
  Week 20: >=75% improvement | 93.6 | 92.4
  Week 20: >=50% improvement | 97.6 | 95.1
  Week 24: 100% improvement | 54.7 | 50.4
  Week 24: >=90% improvement | 83.1 | 78.2
  Week 24: >=75% improvement | 94.2 | 90.3
  Week 24: >=50% improvement | 97.8 | 93.0
  Week 28: 100% improvement | 57.1 | 51.0
  Week 28: >=90% improvement | 85.4 | 77.2
  Week 28: >=75% improvement | 94.0 | 90.3
  Week 28: >=50% improvement | 97.2 | 93.0
  Week 32: 100% improvement | 57.5 | 50.2
  Week 32:>=90 % improvement | 84.8 | 77.4
  Week 32: >=75% improvement | 94.0 | 89.3
  Week 32: >=50% improvement | 97.0 | 93.0
  Week 36: 100% improvement | 58.6 | 50.0
  Week 36: >=90% improvement | 84.5 | 75.7
  Week 36: >=75% improvement | 93.6 | 87.0
  Week 36: >=50% improvement | 97.2 | 92.2
  Week 40: 100% improvement | 58.2 | 48.6
  Week 40: >=90% improvement | 84.6 | 73.7
  Week 40: >=75% improvement | 92.9 | 85.8
  Week 40: >=50% improvement | 95.9 | 90.9
  Week 44: 100% improvement | 58.6 | 49.4
  Week 44: >=90% improvement | 84.1 | 72.6
  Week 44: >=75% improvement | 92.3 | 85.2
  Week 44: >=50% improvement | 94.2 | 91.4
  Week 48: 100% improvement | 58.2 | 48.4
  Week 48: >=90% improvement | 84.5 | 70.0
  Week 48: >=75% improvement | 92.1 | 83.5
  Week 48: >=50% improvement | 94.0 | 89.3
  Week 56: 100% improvement | 50.4 | 27.0
  Week 56: >=90% improvement | 77.3 | 51.4
  Week 56: >=75% improvement | 88.0 | 70.4
  Week 56: >=50% improvement | 91.0 | 82.1

17. Secondary Outcome: Percentage of Participants With IGA Responses Through Week 56
Description: as for outcome 6
Time Frame: Week 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 56
Population: Full analysis set included all the participants randomized at Week 0. Participants who met treatment failure criteria or who had missing IGA score were considered as non-responders for the specific visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percentage of participants
  Week 1: cleared (0) | 0 | 0
  Week 1: cleared (0) or minimal (1) | 3.4 | 2.5
  Week 1: mild or better (=<2) | 27.2 | 34.2
  Week 2: cleared (0) | 0.2 | 0.8
  Week 2: cleared (0) or minimal (1) | 12.4 | 20.2
  Week 2: mild or better (=<2) | 54.1 | 63.8
  Week 3: cleared (0) | 2.6 | 3.3
  Week 3: cleared (0) or minimal (1) | 27.2 | 39.9
  Week 3: mild or better (=<2) | 75.3 | 82.5
  Week 4: cleared (0) | 6.7 | 9.7
  Week 4: cleared (0) or minimal (1) | 44.2 | 59.3
  Week 4: mild or better (=<2) | 85.6 | 92.2
  Week 8: cleared (0) | 29.2 | 35.8
  Week 8: cleared (0) or minimal (1) | 76.6 | 83.5
  Week 8: mild or better (=<2) | 96.3 | 96.3
  Week 12: cleared (0) | 46.3 | 50.2
  Week 12: cleared (0) or minimal (1) | 85.6 | 86.4
  Week 12: mild or better (=<2) | 96.8 | 95.3
  Week 16: cleared (0) | 55.4 | 53.5
  Week 16: mild or better (=<2) | 96.8 | 94.7
  Week 16: cleared (0) or minimal (1) | 86.7 | 86.6
  Week 20: cleared (0) | 56.9 | 53.9
  Week 20: cleared (0) or minimal (1) | 87.8 | 85.6
  Week 20: mild or better (=<2) | 95.3 | 93.2
  Week 24: cleared (0) | 61.0 | 56.0
  Week 24: cleared (0) or minimal (1) | 88.6 | 82.7
  Week 24: mild or better (=<2) | 96.3 | 91.6
  Week 28: cleared (0) | 62.2 | 56.2
  Week 28: cleared (0) or minimal (1) | 87.8 | 82.9
  Week 28: mild or better (<=2) | 95.5 | 90.9
  Week 32: cleared (0) | 63.1 | 54.5
  Week 32: cleared (0) or minimal (1) | 88.6 | 81.5
  Week 32: mild or better (=<2) | 95.5 | 90.5
  Week 36: cleared (0) | 60.7 | 53.7
  Week 36: cleared (0) or minimal (1) | 86.5 | 79.6
  Week 36: mild or better (=<2) | 95.5 | 88.9
  Week 40: cleared (0) | 63.1 | 52.3
  Week 40: cleared (0) or minimal (1) | 86.3 | 78.0
  Week 40: mild or better (=<2) | 93.6 | 87.9
  Week 44: cleared (0) | 62.2 | 51.9
  Week 44: cleared (0) or minimal (1) | 86.0 | 76.5
  Week 44: mild or better (=<2) | 92.3 | 87.5
  Week 48: cleared (0) | 62.2 | 50.4
  Week 48: cleared (0) or minimal (1) | 85.0 | 74.9
  Week 48: mild or better (=<2) | 92.7 | 86.8
  Week 56: cleared (0) | 54.3 | 29.4
  Week 56: cleared (0) or minimal (1) | 78.8 | 58.2
  Week 56: mild or better (=<2) | 87.5 | 76.3

18. Secondary Outcome: Percent Improvement From Baseline in PASI Through Week 56
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72. A higher score indicates more severe disease.
Time Frame: Week 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and Week 56
Population: Full analysis set included all the participants randomized at Week 0. Here 'n' signifies the number of participants analyzed at specified point. Zero percent improvement was assigned from the point when participants met treatment failure criteria and no other data imputation was applied.
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
Number analyzed (Participants) | 534 | 514
Percent improvement
  Week 1: number analyzed (Participants) | 531 | 510
  Week 1 | 20.30 (20.743) | 24.72 (20.711)
  Week 2: number analyzed (Participants) | 533 | 509
  Week 2 | 37.85 (23.567) | 44.56 (23.600)
  Week 3: number analyzed (Participants) | 531 | 507
  Week 3 | 52.76 (24.186) | 60.57 (21.871)
  Week 4: number analyzed (Participants) | 531 | 507
  Week 4 | 64.63 (22.862) | 72.80 (19.478)
  Week 8: number analyzed (Participants) | 531 | 506
  Week 8 | 84.36 (17.278) | 89.40 (13.579)
  Week 12: number analyzed (Participants) | 527 | 505
  Week 12 | 90.85 (14.484) | 92.60 (13.703)
  Week 16: number analyzed (Participants) | 526 | 501
  Week 16 | 93.65 (12.849) | 93.94 (12.123)
  Week 20: number analyzed (Participants) | 525 | 495
  Week 20 | 94.35 (11.525) | 94.41 (12.152)
  Week 24: number analyzed (Participants) | 525 | 490
  Week 24 | 95.27 (9.848) | 93.75 (14.314)
  Week 28: number analyzed (Participants) | 521 | 492
  Week 28 | 95.58 (9.663) | 92.96 (16.835)
  Week 32: number analyzed (Participants) | 521 | 491
  Week 32 | 95.74 (9.336) | 92.95 (16.641)
  Week 36: number analyzed (Participants) | 523 | 487
  Week 36 | 95.45 (11.119) | 92.40 (17.125)
  Week 40: number analyzed (Participants) | 516 | 484
  Week 40 | 95.78 (10.456) | 91.77 (17.733)
  Week 44: number analyzed (Participants) | 511 | 486
  Week 44 | 95.45 (12.293) | 91.34 (18.246)
  Week 48: number analyzed (Participants) | 508 | 478
  Week 48 | 95.76 (11.629) | 90.87 (19.181)
  Week 56: number analyzed (Participants) | 499 | 469
  Week 56 | 93.35 (16.116) | 81.67 (27.627)

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: Safety analysis set included all randomized and treated participants who received at least 1 dose of study agent (partial or complete) at Week 0 according to the actual treatment received during the study.
Arm/Group | Guselkumab 100 mg + Placebo | Secukinumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/534 | 0/511
Serious Adverse Events (participants affected / at risk) | 33/534 | 37/511
Other Adverse Events (participants affected / at risk) | 249/534 | 254/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guselkumab 100 mg + Placebo (N=534) | Secukinumab 300 mg (N=511)
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 1 | 0
Macular Fibrosis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Leukoplakia Oral (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Exercise Tolerance Decreased (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 1
Anaphylactoid Reaction (Immune system disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Neuroborreliosis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram Repolarisation Abnormality (Investigations) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Mixed Anxiety and Depressive Disorder (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Bartholin's Cyst (Reproductive system and breast disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0
Finger Amputation (Surgical and medical procedures) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guselkumab 100 mg + Placebo (N=534) | Secukinumab 300 mg (N=511)
Diarrhoea (Gastrointestinal disorders) | 27 | 20
Nasopharyngitis (Infections and infestations) | 118 | 125
Upper Respiratory Tract Infection (Infections and infestations) | 83 | 92
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 29 | 18
Headache (Nervous system disorders) | 48 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03090100/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03090100/SAP_001.pdf